CLINICAL TRIAL: NCT02853747
Title: Exercise and Arterial Modulation in Youth
Acronym: ExAMIN YOUTH
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Henner Hanssen, Prof.Dr.med. Henner Hanssen, University of Basel
Other Study IDs: EKNZ258/12
Record Dates: First submitted 2016-07-25; First posted 2016-08-03 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Disease; Childhood Obesity; Hypertension; Endothelial Dysfunction
Keywords: arterial stiffness; retinal vessels; physical activity; children
MeSH Terms: conditions — Cardiovascular Diseases; Pediatric Obesity; Hypertension; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Physical Activity, 20-meter shuttle run — cross-sectional physical activity assessment and medical screeening

SUMMARY:
The project is designed as a large scale, cross-sectional study. The aim of the study is to investigate the association of micro- and macrovascular function with physical fitness and body composition in primary school children.

DETAILED DESCRIPTION:
The investigators will examine whether physical fitness, body composition and blood pressure differently affect large and small arteries in young children. Furthermore, the investigators will examine whether pulmonary dysfunction is associated with vascular disorders and if subcutaneous advanced glycation endproducts (AGE's) mediate some of the vascular alterations observed.

ELIGIBILITY:
Inclusion Criteria:

* primary school children aged 6-8 years who can participate in physical education lessons with written consent from their parents.

Exclusion Criteria:

* children with a medical certificate that prohibits physical exercise with no consent from their parents.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ExAMIN YOUTH is a cooperative project between the department of sport, movement and health sciences (DSBG) of the University of Basel and the Cantonal Office of Sport of Basel-Stadt (COS-BS). Primary school children aged 6 to 8 years of the City of Basel are examined.The investigators expect to include n=1200 children in this cross-sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Association of arterial stiffness (pulse wave velocity) with physical fitness in primary school children | Through study completion, an average of 1 year.
  Oscillometric calculation of central pulse wave velocity.

SECONDARY OUTCOMES:
Association of arteriolar-to-venular diameter ratio (AVR) with physical fitness in primary school children | Through study completion, an average of 1 year.
  Retinal vessel diameters by use of Static Retinal Vessel Analyzer (SVA-T).
Association of subcutaneous advanced glycation endproducts (AGEs) with body composition, blood pressure and physical fitness | Through study completion, an average of one year.
  Non-invasive, subcutaneous measurement of AGEs (skin autofluorescence).
Association of lung function (FEV1/VC) with body composition, blood pressure and physical fitness | Through study completion, an average of one year.
  Handheld spirometer (EasyOne Diagnostic) to measure vital capacity (VC), peak expiratory flow (PEF), forced expiratory volume (FEV1) and the ratio of FEV1/VC.

CONTACTS AND LOCATIONS:
Overall Officials: Henner Hanssen, Prof. Dr. med., Principal Investigator — University of Basel; Lukas Zahner, Prof. Dr., Principal Investigator — University of Basel
Locations (1):
- Bereich Sport- und Bewegungsmedizin, Abteilung Präventive Sportmedizin und Systemphysiologie, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Imhof K, Zahner L, Schmidt-Trucksass A, Faude O, Hanssen H. Influence of physical fitness and activity behavior on retinal vessel diameters in primary schoolchildren. Scand J Med Sci Sports. 2016 Jul;26(7):731-8. doi: 10.1111/sms.12499. Epub 2015 Jun 24. PMID 26105148
- [Background] Veijalainen A, Tompuri T, Haapala EA, Viitasalo A, Lintu N, Vaisto J, Laitinen T, Lindi V, Lakka TA. Associations of cardiorespiratory fitness, physical activity, and adiposity with arterial stiffness in children. Scand J Med Sci Sports. 2016 Aug;26(8):943-50. doi: 10.1111/sms.12523. Epub 2015 Jul 29. PMID 26220100
- [Background] Steinmann M, Abbas C, Singer F, Casaulta C, Regamey N, Haffner D, Fischer DC, Simonetti GD. Arterial stiffness is increased in asthmatic children. Eur J Pediatr. 2015 Apr;174(4):519-23. doi: 10.1007/s00431-014-2423-2. Epub 2014 Sep 25. PMID 25248341
- [Derived] Hauser C, Lichtenstein E, Nebiker L, Streese L, Kochli S, Infanger D, Faude O, Hanssen H. Cardiorespiratory fitness and development of childhood cardiovascular risk: The EXAMIN YOUTH follow-up study. Front Physiol. 2023 Aug 23;14:1243434. doi: 10.3389/fphys.2023.1243434. eCollection 2023. PMID 37680774
- [Derived] Kochli S, Smith W, Lona G, Goikoetxea-Sotelo G, Breet Y, Botha-Le Roux S, Mokwatsi GG, Kruger R, Hanssen H. Obesity, blood pressure and retinal microvascular phenotype in a bi-ethnic cohort of young children. Atherosclerosis. 2022 Jun;350:51-57. doi: 10.1016/j.atherosclerosis.2022.04.018. Epub 2022 Apr 21. PMID 35490596
- [Derived] Kochli S, Deiseroth A, Hauser C, Streese L, Schmidt-Trucksass A, Faude O, Hanssen H. Body Composition and Physical Fitness Affect Central Hemodynamics in Young Children. Front Pediatr. 2021 Oct 27;9:750398. doi: 10.3389/fped.2021.750398. eCollection 2021. PMID 34778141
- [Derived] Kochli S, Endes K, Grenacher J, Streese L, Lona G, Hauser C, Deiseroth A, Zahner L, Hanssen H. Socioeconomic Status and Parental Lifestyle Are Associated With Vascular Phenotype in Children. Front Public Health. 2021 Mar 26;9:610268. doi: 10.3389/fpubh.2021.610268. eCollection 2021. PMID 33842418
- [Derived] Kochli S, Endes K, Bartenstein T, Usemann J, Schmidt-Trucksass A, Frey U, Zahner L, Hanssen H. Lung function, obesity and physical fitness in young children: The EXAMIN YOUTH study. Respir Med. 2019 Nov;159:105813. doi: 10.1016/j.rmed.2019.105813. Epub 2019 Nov 8. PMID 31731085
- [Derived] Kochli S, Endes K, Steiner R, Engler L, Infanger D, Schmidt-Trucksass A, Zahner L, Hanssen H. Obesity, High Blood Pressure, and Physical Activity Determine Vascular Phenotype in Young Children. Hypertension. 2019 Jan;73(1):153-161. doi: 10.1161/HYPERTENSIONAHA.118.11872. PMID 30571553